CLINICAL TRIAL: NCT03088514
Title: Investigation of Dietary Nitrate Effects in Hypertension-induced Target Organ Damage
Acronym: NITRATE-TOD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Collaborators: Barts & The London NHS Trust (Other)
Responsible Party: Principal Investigator, Amrita Ahluwalia, Professor of Vascular Pharmacology, Queen Mary University of London
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 10/H0703/98
Record Dates: First submitted 2017-03-09; First posted 2017-03-23 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Hypertension
Keywords: Hypertension; Left Ventricular Hypertrophy; Endothelial Dysfunction; Nitrate
MeSH Terms: conditions — Hypertension; Hypertrophy, Left Ventricular

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- NITRATE-LVH intervention (Experimental): 70ml of beetroot juice (approximately 6-8 mmol of inorganic nitrate) once a day for 4 months
  Interventions: Dietary Supplement: Beetroot juice
- NITRATE-LVH placebo (Placebo Comparator): 70ml of beetroot juice (no inorganic nitrate) once a day for 4 months
  Interventions: Dietary Supplement: Beetroot juice
- NITRATE-CBP intervention (Experimental): 70ml of beetroot juice (approximately 6-8 mmol of inorganic nitrate) once a day for 4 month
  Interventions: Dietary Supplement: Beetroot juice
- NITRATE-CBP placebo (Placebo Comparator): 70ml of beetroot juice (no inorganic nitrate) once a day for 4 months
  Interventions: Dietary Supplement: Beetroot juice

INTERVENTIONS:
Dietary Supplement: Beetroot juice — Beetroot juice (70ml daily) with or without inorganic nitrate

SUMMARY:
This study aims to determine whether dietary inorganic nitrate (in beetroot juice) is able to reduce overall thickening of the heart (left ventricular hypertrophy or LVH) and stiffness of the arteries when given to patients with persistently raised blood pressure (hypertension). Half the patients will receive the beetroot juice containing inorganic nitrate and half will receive beetroot juice from which the inorganic nitrate has been removed. The volunteers will take the juice every day for 4 months.

DETAILED DESCRIPTION:
In hypertension persistent raised blood pressure (BP) is associated with endothelial dysfunction, arterial stiffness and left ventricular (LV) remodeling that are key phenomena associated with the pathogenesis and complications of hypertension.

One of the main substances that the healthy endothelium produces that is responsible for maintaining the patency of blood vessels is nitric oxide (NO). In hypertension, one of the key pathogenic effects is the dysfunction of the endothelium characterized by a decrease in ability to generate nitric oxide (NO). Previous studies have shown that dietary inorganic nitrate supplementation lowers blood pressure (Kapil et al. 2015), however, whether this approach might also improve endothelial function and LV remodeling is unknown. The effects of inorganic nitrate are due to its conversion in the body to inorganic nitrite and thereafter to NO.

This study will assess the effects of dietary inorganic nitrate on LVH using cardiac magnetic resonance imaging (NITRATE-LVH arm). In addition, the effects of dietary inorganic nitrate on central aortic blood pressure, arterial stiffness using pulse wave velocity and endothelial function using flow mediated dilatation will be evaluated (NITRATE-CBP arm).

ELIGIBILITY:
Inclusion Criteria:

1. Patients will be enrolled following an informed consent. The subject will be able to understand and comply with protocol requirements, instructions and protocol restrictions.
2. Aged 18-80 years.
3. The study subjects will be hypertensives with evidence of difficulty treating to target BP (daytime ABPM 135-170/85-105 mmHg) on 1 or more antihypertensive agents, with insufficient efficacy or intolerance of medications.
4. For NITRATE LVH, echocardiographic evidence of LV hypertrophy (LV mass indexed to body surface area (BSA); males >115g/m2; females >95 g/m2).
5. Patients will have been established on an antihypertensive treatment regime for at least 1 month by the time of participation in the study and will not require changes in pharmacological intervention for the duration of the trial.

Exclusion Criteria:

Unless specified, a subject will not be eligible for inclusion in this study if any of the following criteria apply:

1. History of chronic viral hepatitis (including presence of hepatitis B surface antigen or hepatitis C antibody), or other chronic hepatic disorders.
2. History of increased liver function tests (ALT, AST) due to acute or chronic liver conditions, 3x above the upper limit of normal or bilirubin 1.5x above the upper limit of normal at screening.
3. Renal impairment with creatinine clearance (eGFR) of <50 ml/min at screening.
4. Patients with diabetes mellitus, defined by previous history of diabetes or HbA1c >6.5% (>48 mmol/mol) at screening.
5. Subjects with LDLc, >7.5 mmol/l. TG level >10mmol/l.
6. History of heart failure defined as NYHA class II - IV or those with known LV dysfunction (EF<40%) regardless of symptomatic status
7. History of malignancy within the past 5 years, other than non-melanoma skin cancer.
8. Current life-threatening condition other than vascular disease (e.g. very severe chronic airways disease, HIV positive, life-threatening arrhythmias) that may prevent a subject from completing the study.
9. Use of an investigational device or investigational drug within 30 days or 5 half-lives (whichever is longer) preceding the first dose of study medication.
10. Subjects who will commence or who are likely to commence regular treatment with non-steroidal anti-inflammatory drugs (NSAIDs) (other than aspirin), from screening until study completion.
11. Any non-stable dosing of ongoing medication regimens throughout the study trial.
12. Drug abuse within the past 6 months.
13. The subject has a three-month prior history of regular alcohol consumption exceeding an average weekly intake of > 28 units (or an average daily intake of greater than 3 units) for males, or an average weekly intake of > 21 units (or an average daily intake of greater than 2 units) for females. 1 unit is equivalent to a half-pint (284mL) of beer/lager; 25mL measure of spirits or 125mL of wine.
14. Any other subject whom the Investigator deems unsuitable for the study (e.g. due to other medical reasons, laboratory abnormalities, expected study medication noncompliance, or subject's unwillingness to comply with all study-related study procedures).
15. Subjects with rheumatoid arthritis, connective tissue disorders and other conditions known to be associated with chronic inflammation (e.g. Inflammatory Bowel Disease).
16. Subjects with any acute infection, or recent systemic (oral or IV) antibiotics within 1 month of screening, or significant trauma (burns, fractures).
17. Subjects who have donated more than 500 mL of blood within 56 days prior to the study medication administration.
18. Self reported use of anti-microbial mouthwash or tongue scrapes.
19. Concomitant xanthine oxidase inhibitors (such as allopurinol).
20. Known history of significant claustrophobia, previous intolerance of CMR imaging or known (or suspected) incompatible metallic implant.
21. Pregnancy.
22. Allergy to gadolinium-based contrast agents used for CMR.
23. Patients with known LVH caused by another established pathology diagnosed prior to or at screening e.g. severe aortic stenosis, hypertrophic cardiomyopathy, amyloidosis and Fabry's disease.

Exceptions to the exclusion criteria:

* For criteria 18, patients can enter the trial if they discontinue the use of anti-microbial mouthwash for the duration of the clinical trial.
* nCriteria 20 and 22 do not apply to participants who will not have a CMR scan in the NITRATE-CBP arm

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2017-03-23 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2023-11-15 (Actual)

PRIMARY OUTCOMES:
Left ventricular hypertrophy regression | 4 months
  change in LV mass as assessed using cardiac magnetic resonance imaging
Pulse wave velocity | 4 months
  non-invasive measures of arterial stiffness
Central blood pressure | 4 months
  non-invasive measure of central blood pressure

SECONDARY OUTCOMES:
Flow mediated dilatation (FMD) | 4 months
  non-invasive measure of endothelial function using ultrasound
Brachial blood pressure | 4 months
  brachial blood pressure
Change in plasma nitrate levels | 4 months
  assessed by chemiluminescence
Change in plasma nitrite levels | 4 months
  assessed by chemiluminescence
Change in nitric oxide activity (cGMP) | 4 months
  nitric oxide activity measured by determining plasma concentrations of cyclic guanosine monophosphate (cGMP)

CONTACTS AND LOCATIONS:
Overall Officials: Amrita Ahulwalia, BSc PhD, Principal Investigator — Queen Mary University of London
Locations (1):
- Queen Mary University of London, London, United Kingdom

REFERENCES:
- [Background] Kapil V, Khambata RS, Robertson A, Caulfield MJ, Ahluwalia A. Dietary nitrate provides sustained blood pressure lowering in hypertensive patients: a randomized, phase 2, double-blind, placebo-controlled study. Hypertension. 2015 Feb;65(2):320-7. doi: 10.1161/HYPERTENSIONAHA.114.04675. Epub 2014 Nov 24. PMID 25421976
- [Derived] Lau CWZ, Hamers AJP, Rathod KS, Shabbir A, Cooper J, Primus CP, Davies C, Mathur A, Moon JC, Kapil V, Ahluwalia A. Randomised, double-blind, placebo-controlled clinical trial investigating the effects of inorganic nitrate in hypertension-induced target organ damage: protocol of the NITRATE-TOD study in the UK. BMJ Open. 2020 Jan 21;10(1):e034399. doi: 10.1136/bmjopen-2019-034399. PMID 31969369